CLINICAL TRIAL: NCT02239406
Title: Acetabular Bone Vascularity in Metal-on-Metal Revisions
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment interest.
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Presbyterian Pathology Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: HK025
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Failure of Total Hip
Keywords: metal on metal total hip; avasuclar necrosis; acetabular revision; bone vascularity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Metal-on-Metal Revision: Patients who have a failed metal on metal total hip implant and are presenting for revision surgery

SUMMARY:
The purpose of this study is to determine if avascular necrosis of the acetabulum is present in metal-on-metal revisions and to what depth this dead avascular bone occurs.

A convenient sample of a consecutive series of 15 patients treated for metal on metal acetabular revision surgery will be included.

DETAILED DESCRIPTION:
Patients being treated for metal on metal acetabular revision surgery by a physician at OrthoCarolina, PA will be screened for eligibility. These patients will be approached by their surgeon and asked to volunteer their participation in the study. Potential subjects will meet with a research coordinator to discuss details of the study and those you volunteer participation will be asked to sign an informed consent prior to the collection of study data. . Basic demographic information (initials, age, gender, height, weight, BMI), dates of original index surgery, reason for revision, type of implant being removed, and standard of care cobalt and chromium metal ion levels will be collected via chart review.

Patients who meet all eligibility criteria will have three biopsies performed at the time of their revision surgery. A pathologist will note the presence or absence of bone necrosis and will measure the length (mm) of necrosis, acute inflammation, chronic inflammation, normal bone, and entire bone specimen in order to obtain a ratio.

Biopsy Protocol:

A bone biopsy is a procedure in which bone samples are removed (with a special instrument during surgery) and looked at under a microscope for necrosis (tissue death), infection, or other bone disorders. Once the acetabular hip replacement implants have been removed the following steps will occur:

* The biopsy needle will be inserted into the bone (3 locations; 2 from ilium, 1 from pubis or ischium = 3 total).
* The biopsy needle will be withdrawn and firm pressure will be applied to the biopsy site for a few minutes, until the bleeding has stopped.
* Each bone biopsy sample will be labeled sequentially and by anatomic location (i.e., ilium #1, ilium #2)
* The normal bone will be marked on the bone sample.
* The bone biopsy sample will be sent to the lab for examination.
* The acetabulum bone will be reamed so the new implant can be seated.

ELIGIBILITY:
Inclusion Criteria:

* Patients being revised for an aseptic metal on metal acetabular revision.
* Patient is greater than one year postoperative.
* Patient has had cobalt and chromium metal ion levels tested within 6 months of the planned revision surgery.
* Understands the local language and is willing and able to follow the requirements of the protocol.
* Understands the informed consent and signs the institutional review board or independent ethics committee (IRB/IEC) approved informed consent form.

Exclusion Criteria:

* History of infection
* Evidence of current substance or alcohol abuse
* Being treated with radiation, chemotherapy, immunosupression, or chronic steroid therapy (prednisone use up to 5 mg/qd or its equivalent is allowed)
* Is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of a total of 15 patients will be enrolled at OrthoCarolina.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The depth (mm) of avascular bone from the acetabular surface per each patient | participants will be followed for the duration of their surgery, an expected average of 2 hours
  A bone biopsy is a procedure in which bone samples are removed (with a special instrument during surgery) and looked at under a microscope for necrosis (tissue death), infection, or other bone disorders. Once the acetabular hip replacement implants have been removed the following steps will occur:
  * The biopsy needle will be inserted into the bone (3 locations; 2 from ilium, 1 from pubis or ischium = 3 total).
  * The biopsy needle will be withdrawn and firm pressure will be applied to the biopsy site for a few minutes, until the bleeding has stopped.
  * Each bone biopsy sample will be labeled sequentially and by anatomic location (i.e., ilium #1, ilium #2)
  * The normal bone will be marked on the bone sample.
  * The bone biopsy sample will be sent to the lab for examination.

SECONDARY OUTCOMES:
The ratio of necrotic bone per each patient | paricipants will be followed for the duration of their surgery, an expected average of 2 hours
  The ratio of each bone type (necrotic, acute inflammation, chronic inflammation, and normal bone) in relation to the length of the entire bone specimen will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fehring, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No